CLINICAL TRIAL: NCT01748500
Title: Pantoprazole and Docetaxel for Men With Metastatic Castration-Resistant Prostate Cancer - a Single Arm Phase II Clinical Trial With a Predefined Reference Group (PANDORA)
Brief Title: Pantoprazole and Docetaxel for Men With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANDORA; 12-0388-C (Other: UHN REB)
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
Keywords: metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pantoprazole, Docetaxel, Prednisone (Experimental)
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole
  Other Names: Pantoprazole sodium

SUMMARY:
The main objectives of this trial are:

1. To assess the activity and safety of pantoprazole and docetaxel (with prednisone) in men with metastatic CRPC who have not received prior chemotherapy.
2. To evaluate archival prostate cancer tissue of men included in the clinical trial for evidence of autophagy using IHC for LC3B, ATG5, p62 as well as ERG.
3. To evaluate pharmacokinetic interactions of pantoprazole with docetaxel.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18yrs
* ECOG performance status ≤2
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Clinical or radiological evidence of metastatic disease
* Disease progression while receiving androgen deprivation therapy with an increase in PSA of 25% or greater over nadir value measured on 3 consecutive occasions at least 1 week apart
* Antiandrogen therapy must have been stopped at least 4 weeks prior to start of trial treatment (6 weeks in the case of bicalutamide or nilutamide)if there was a reduction in serum PSA after this therapy was initiated
* Baseline serum prostate-specific antigen (PSA)≥10ng/ml
* Total testosterone <50 ng/dL (<1.7 nmol/L)
* Adequate hematologic values: neutrophil count ≥1,500/mm3, platelet ≥100,000/mm3, hemoglobin ≥10.0 g/dl
* Adequate hepatic and renal function: total bilirubin level ≤1.5 x ULN (unless secondary to documented Gilbert's disease); ALT,AST, and creatinine ≤1.5 x ULN
* Ability to understand and to sign consent for the study

Exclusion Criteria:

* Prior treatment for prostate cancer with chemotherapy or radioisotopes
* History of another cancer within the preceding five years (except basal or squamous-cell skin cancer or adequately treated superficial bladder cancer)
* Known or suspected brain or leptomeningeal metastases
* Symptomatic peripheral neuropathy of grade 2 or higher
* Major surgery within 4 weeks of start of trial treatment
* Radiotherapy to ≥25% of the bone marrow and any radiotherapy within 4 weeks of start of trial treatment
* Known hypersensitivity to trial treatment or hypersensitivity to any of its components
* Any concomitant drugs contraindicated for use with the trial treatment
* Any serious underlying medical condition which could impair the ability of the patient to participate in the trial
* Any psychological, familial, sociological or other patient related factors that might preclude compliance with the study protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-01; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Confirmed PSA response | 20 months
  The primary endpoint is met if PSA falls to ≤50% of baseline, maintained for ≥3 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada